CLINICAL TRIAL: NCT03213730
Title: Perceptual-Cognitive Training After a Mild Traumatic Brain Injury: Towards a Sensitive Marker for Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Isabelle Gagnon, Clinical Scientist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-146-PED
Record Dates: First submitted 2017-07-09; First posted 2017-07-11 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Brain Concussion; Post-Concussion Symptoms; Concussion
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Standard care + 3D-MOT protocol.
  Interventions: Other: 3D-MOT Neurotracker
- Active control group (Active Comparator): Standard care + visual attention task (2048 online game)
  Interventions: Other: Visual Attention Intervention
- Control group (No Intervention): Standard care alone

INTERVENTIONS:
Other: 3D-MOT Neurotracker — A predetermined number of spheres (eight) are presented in the 3D-MOT task. The spheres are all identical in shape and color. Before each trial, four spheres are highlighted, and then returned to their original color. Participants will be asked to track those four spheres for the duration of the trial (8 seconds). Spheres will be moving, bouncing, colliding, until they finally stop moving and the participant has to identify the spheres that were initially highlighted. Previous work with healthy individuals has shown that the minimum optimal number of sessions (3 blocks) necessary to induce brain plasticity and enhance other, "non-trained" brain functions is between 5-6. The training protocol will therefore include 6 sessions (3 blocks each), at intervals of 48 to 72 hours, over a maximum of 3 weeks.
  Arms: Experimental group
Other: Visual Attention Intervention — The visual attention intervention will consist of the 2048 game, a single-player sliding block puzzle game of which the objective is to slide numbered tiles on a grid to combine them to create number 2048. 2048 is played on a gray 4×4 grid, with numbered tiles that slide smoothly when a player moves them using the four arrow keys. Every turn, a new tile will randomly appear in an empty spot on the board with a value of either 2 or 4.Tiles slide as far as possible in the chosen direction until they are stopped by either another tile or the edge of the grid. If two tiles of the same number collide while moving, they will merge into a tile with the total value of the two tiles that collided. Higher-scoring tiles emit a soft glow. Children will play for a time equivalent to that of the 3D-MOT.
  Arms: Active control group

SUMMARY:
This study is part of a larger, multi-centered project done with the collaboration of University Of Victoria. This study holds three separate studies on the mild traumatic brain injured population and the use of perceptual-cognitive training (3D-MOT).

ELIGIBILITY:
Inclusion Criteria:

* The child experienced a head injury (a direct or indirect blow to the head) resulting in concussion-like symptoms (e.g. headache, nausea, balance problems, tiredness, visual problems, cognitive issues) in the previous 72 hours
* Parent/legal guardian speak English or French
* The child speak English or French

Exclusion Criteria:

* Previous concussion in the last 6 months, or any previous concussion with unresolved symptoms
* Multi-system injuries requiring admission, operating room, procedural sedation in the Emergency Department
* Other co-existing injuries, co-morbidities or diagnoses preventing participation to intervention/assessment of gait and balance
* Pre-morbid or co-morbid condition affecting visual function
* Patient intoxicated at the time of injury
* Significant developmental delay
* Loss of consciousness prior to head injury

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Post Concussion Symptom Inventory | 1 month
  Post-concussion symptoms checklist

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Children's Hospital, MUHC, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Teel E, Brossard-Racine M, Corbin-Berrigan LA, Gagnon I. Perceptual Cognitive Training Does Not Improve Clinical Outcomes at 4 and 12 Weeks Following Concussion in Children and Adolescents: A Randomized Controlled Trial. J Head Trauma Rehabil. 2021 Mar-Apr 01;36(2):E97-E107. doi: 10.1097/HTR.0000000000000633. PMID 33201041